CLINICAL TRIAL: NCT05658172
Title: SURVIVE (Standard Surveillance vs. Intensive Surveillance in Early Breast Cancer) - a Partially Double-blinded, Multi-center, Randomized, Controlled Superiority Study
Brief Title: Standard Surveillance vs. Intensive Surveillance in Early Breast Cancer
Acronym: SURVIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Wolfgang Janni (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor-Investigator, Prof. Wolfgang Janni, Director of the clinic for gynecology and obstetrics, University of Ulm
Organization: University of Ulm (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: SURVIVE; 01KD2202 (Other Grant/Funding Number: German Federal Ministry of Education and Research (BMBF)); DRKS00030745 (Registry Identifier: Deutsches Register Klinischer Studien (DRKS))
Record Dates: First submitted 2022-11-23; First posted 2022-12-20 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
Keywords: medium risk; high risk
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a partially double-blinded, multi-center, randomized, controlled superiority study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study will be performed as partially double-blinded. This means, all patients and doctors are blinded initially as blood sampling is done in all patients, irrespective of randomization to the Standard Surveillance arm or the Intensive Surveillance arm. If one of the biomarkers (CA27.29, CEA, CA125, CTC, ctDNA) is abnormal and requires a confirmatory blood sampling or triggers imaging, unblinding is the consequence as these patients will be asked to undergo further assessments and the responsible doctor will arrange these. Unblinding in this case is the ethical consequence of not letting all patients undergo a confirmatory blood sampling or even undergo additional imaging without elevated biomarkers. If no confirmatory blood sampling or imaging is necessary, patients in the Intensive Surveillance arm will not be unblinded as there is no purpose to serve. Patients in the Standard Surveillance arm will not be unblinded altogether.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Surveillance arm (Active Comparator): Intensified surveillance. Prospective tumor marker (CA27.29, CA125, CEA), CTC and ctDNA testing of the blood samples. Abnormal findings of either marker (CA27.29 and/or CA125 and/or CEA and/or CTC and/or ctDNA) will be regarded as molecular relapse and trigger diagnostic imaging.
  Interventions: Diagnostic Test: Determination of tumormarkers (CA27.29, CEA, CA125); Diagnostic Test: Determination of CTC levels; Diagnostic Test: Determination of ctDNA levels
- Standard Surveillance arm (Placebo Comparator): Surveillance according to national guidelines. Blood samples will not be analyzed immediately and will therefore not trigger imaging. A biobank will be established for retrospective and translational studies. This procedure is necessary to ensure the partially double-blinded study design.
  Interventions: Other: Biobanking of blood samples

INTERVENTIONS:
Diagnostic Test: Determination of tumormarkers (CA27.29, CEA, CA125) — CA27.29, CEA and CA125 will be measured with the AIA®-CL1200 by TOSOH BIOSCIENCE (TOSOH CORPORATION, Tokyo, Japan). The CL AIA-PACK assays are two-step chemiluminescence enzyme immunoassay kits. CA27.29/CEA/CA125 present in a test sample is bound to the anti- CA27.29/CEA/CA125 mouse monoclonal antibody immobilized on the magnetic microparticles in one cell (Cell-I). After first incubation, the magnetic microparticles are washed and the enzyme-labeled anti- CA27.29/CEA/CA125 mouse monoclonal antibody that has been reconstituted in another cell (Cell-II) is dispensed into Cell-I. After second incubation, the magnetic microparticles are washed again and are incubated with a chemiluminescent substrate, DIFURAT®. The amount of enzyme-labeled antibodies that bind to the magnetic microparticles is directly proportional to the CA27.29/CEA/CA125 concentration in the test sample. A standard curve is constructed, unknown sample concentrations are calculated by using this curve.
  Other Names: Chemiluminescence enzyme immunoassay
  Arms: Intensive Surveillance arm
Diagnostic Test: Determination of CTC levels — CTCs will be analyzed using the CellSearch® System (Menarini Silicon Biosystems). The CellSearch® system is designed to enumerate CTCs of epithelial origin (CD45-, EpCAM+, cytokeratin 8+ / 18+ and/or 19+). The basic principle is linking a magnetic ferrofluid reagent that contains i. a. antibodies targeting the EpCAM antigen to CTCs. After steps of immunomagnetic capture and enrichment as well as addition of fluorescent reagents (that contain anti-CK-PE, DAPI and anti-CD45-APC), the automatic dispersion to a magnetic cartridge holder takes place. Via strong magnetic field, the magnetically labeled epithelial cells are attracted to the surface of the cartridge where they can be scanned automatically. Images of events where CK-PE and DAPI fluorescence are co-located are presented to the user for final classification. An event is classified as a tumor cell when its morphological features are consistent with that of a tumor cell and it exhibits the phenotype EpCAM+, CK+, DAPI+ and CD45-.
  Other Names: CellSearch® System
  Arms: Intensive Surveillance arm
Diagnostic Test: Determination of ctDNA levels — Presence of ctDNA will be analyzed centrally at Inivata Inc. using the RaDaRTM assay. Therefore, primary tumor tissue and peripheral blood specimens will be shipped for centralized analysis to Inivata Inc. RaDaRTM is a tumor-informed approach, beginning with whole exome sequencing of a tumor specimen from a patient's biopsy or surgical resection. SNVs and indels identified from the exome sequencing are prioritized to build a patient specific primer panel of up to 48 tumor-specific somatic variants. Patient specific primers are combined with common SNP primers for NGS for quality control purposes. To detect patient specific ctDNA, NGS testing is performed with the RaDaRTM assay using a multiplex PCR based on the InVision® platform.
  Other Names: RaDaRTM assay
  Arms: Intensive Surveillance arm
Other: Biobanking of blood samples — To ensure the possibility of retrospective studies during and after the ongoing study, a biobank will be implemented.
  Other Names: Translational research
  Arms: Standard Surveillance arm

SUMMARY:
The goal of this clinical study is to evaluate the potential benefits of intensified surveillance versus standard surveillance in medium-risk and high-risk early breast cancer patients.

The main questions it aims to answer are:

* Comparison of the 5-year ob´verall survival rates between patients in the Standard Surveillance arm versus patients in the liquid-biopsy guided Intensive Surveillance arm
* Determination of the Overall Lead Time Effect generated due to tumor marker/CTC/ctDNA guided Intensive Surveillance compared to Standard Surveillance after primary therapy in early breast cancer patients.

Participants will recieve regular blood drawals. Solely the blood samples of the intensive surveillance arm will be analysed for prospective tumor markers/CTCs/ctDNAs. Abnormal findings of either marker will trigger diagnostic imaging to search for possible metastases. The blood samples of the standard surveillance arm will solely be biobanked for future research purposes.

DETAILED DESCRIPTION:
This is a partially double-blinded, multi-center, randomized, controlled superiority study to evaluate the potential benefits of intensified surveillance versus standard surveillance in medium-risk and high-risk early breast cancer patients.

3500 patients will be enrolled after completion of primary anti-tumor therapy (adjuvant chemotherapy, surgery or radiotherapy, whichever occurs last) and randomized in a 1:1 ratio to receive:

* Standard Surveillance according to national guidelines or
* Intensive Surveillance with additional testing of blood samples for prospective tumor markers (CA27.29, CA125, CEA), CTC and ctDNA

In both study arms patients will receive standard surveillance according to national guidelines, including clinical follow-up visits every 3 months for the first 3 years and every 6 months for the following 2 years. Additionally, blood samples will be drawn and Quality of Life (QoL) will be analyzed at these clinical follow-up visits in both arms.

In the Standard Surveillance arm blood samples will be stored in a biobank. In the Intensive Surveillance arm blood samples will be tested for prospective tumor markers (CA27.29, CA125, CEA), CTCs and ctDNA. Abnormal findings of either marker (CA27.29 or CA125 or CEA or CTC or ctDNA) will trigger diagnostic imaging. Additionally, blood samples will be stored in a biobank for retrospective analysis.

In both study arms detection of distant recurrence will terminate the surveillance protocol and treatment will be initiated according to national guidelines.

Planned enrollment period is approximately 24 months, total study duration is approximately 144 months (2-year recruitment period, 5-year interventional period, 5-year follow up period). In terms of long-term follow-up after end of study, patients have the possibility to participate in the patient self-reporting registry (Patientenselbstauskunft).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent for all study procedures according to local regulatory requirements prior to beginning specific protocol procedures.
2. Unilateral or bilateral primary invasive carcinoma of the breast, confirmed histologically.
3. Patients with intermediate- to high-risk early breast cancer defined as either

   * an indication for (neo-)adjuvant chemotherapy (regardless whether performed or not), and/or
   * Large tumor (> 50 mm), and/or
   * Positive lymph nodes, and/or
   * High grade (>= G3). Indication to (neo-)adjuvant chemotherapy is seen as stated in the German S3 guideline for breast cancer as well as stated in the guidelines from the AGO.
4. A complete resection of the primary tumor, with resection margins free of invasive carcinoma.
5. Completion of primary anti-tumor therapy (adjuvant chemotherapy, surgery or radiotherapy, whichever occurs last) at least 4 weeks but no more than 24 months previously. Enrollment of patients during any kind of adjuvant therapy except chemotherapy (e.g., but not limited to endocrine therapy, antibody therapy, CDK4/6-inhibitors, PARP inhibitors, PI3K inhibitors, antibody-drug conjugates and other novel agents) is allowed.
6. Availability of primary tumor tissue from core biopsy or surgical removed tissue (FFPE Slide (≥ 6 mm³, min. 10 slides, thickness: 5 µm-10 µm, area >150 mm² and 1 H&E stained slide, minimum 20% tumor content) or FFPE Block (≥ 6 mm³ thickness: 100 µm, area: >150 mm² and 1 H&E stained slide, minimum 20% tumor content) or Genomic DNA extracted from FFPE slides or block (≥ 600 ng, Minimum volume: 25 µL, concentration: 20 ng/µL, buffer: 10 mM Tris pH 8, 1 mM EDTA)) at timepoint of enrollment.

   * Patients with primary systemic therapy: tissue from core biopsy
   * Patients receiving surgery as primary therapy: surgically removed cancer tissue.
7. No current clinical evidence for distant metastases.
8. Females or males ≥ 18 years and ≤ 75 years of age.
9. Performance status ≤ 1, Eastern Cooperative Oncology Group (ECOG) scale.
10. Patient must be willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Patients with a history of any secondary primary malignancy are ineligible with the following exceptions:

   * in situ carcinoma of the cervix or
   * adequately treated basal cell carcinoma of the skin or
   * ipsi- or contralateral non-invasive carcinoma of the breast (DCIS).
2. Patients in pregnancy or breastfeeding. If a patient gets pregnant during the participation in the interventional phase of the study (Year 1-5), an end of intervention visit will be scheduled and the patient will enter the follow-up phase of the study. Pregnancy during the follow-up phase of the study is to be reported but does not lead to an exclusion of the study.
3. History of significant neurological or psychiatric disorders including psychotic disorders, dementia or seizures that would prohibit the understanding and giving of informed consent.
4. Renal insufficiency with GFR < 30 mL/min.
5. Previous or concomitant cytotoxic or other systemic antineoplastic treatment that is not used for treating the primary breast cancer.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3500 (Estimated)
Dates: Start 2022-12-07 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 10 years
  OS is defined as time from randomization until the death of the patient independent of cause of death. If a patient is not known to have died, OS is censored at the date of last contact.
Overall Lead Time Effect | 5 years
  This endpoint is a composite measure, defined as the median time from molecular to via Imaging verified Recurrence Lead Time (calculated only for patients in the liquid-biopsy guided Intensive Surveillance arm) + Difference in time to distant recurrence between the two arms (i.e., difference between median time from randomization to distant recurrence for all patients with distant recurrence in the Standard Surveillance arm and median time from randomization to distant recurrence for all patients with distant recurrence in the liquid-biopsy guided Intensive Surveillance arm). The Overall Lead Time Effect will be assessed for all markers in combination.

SECONDARY OUTCOMES:
Invasive disease-free survival (IDFS) | 10 years
  IDFS is defined as time from randomization until first IDFS event, including any invasive ipsilateral, regional, contralateral, and distant disease recurrence, second primary tumors, or death from any cause as event; non-invasive, in-situ cancer events are excluded. If a patient has not had an event, IDFS is censored at the date of last adequate tumor assessment.
Distant disease-free survival (DDFS) | 10 years
  DDFS is defined as time from randomization until first DDFS event including metastasis, second primary tumors and death from any cause as event. If a patient has not had an event, DDFS is censored at the date of last adequate tumor assessment.
Distant recurrence-free survival (DRFS) | 10 years
  DRFS is defined as time from randomization until first DRFS event including metastasis and second primary tumors; death from any cause is not included as event. If a patient has not had an event, DRFS is censored at the date of last adequate tumor assessment.
Breast cancer specific survival (BCSS) | 10 years
  BCSS is defined as time from randomization until breast cancer associated death of the patient. If a patient is not known to have died, BCSS is censored at the date of last contact. If a patient has died for reasons not associated with breast cancer (by clinical assessment), BCSS is censored at the date of death.
Invasive breast cancer free survival (IBCFS) | 10 years
  IBCFS is defined as time from randomization until first IBCFS event, including any invasive ipsilateral, regional, contralateral and distant disease recurrence or death from any cause as event; non-invasive, in-situ cancer events are excluded. If a patient has not had an event, IBCFS is censored at the date of last adequate tumor assessment.
Overall Survival (OS) after 10 Years | 10 years
  OS is defined as time from randomization until the death of the patient independent of cause of death. If a patient is not known to have died, OS is censored at the date of last contact.
Molecular to via Imaging verified Recurrence Lead Time in the Interventional arm | 5 years
  The Lead Time is defined as time from first molecular relapse to via imaging verified recurrence for all patients in the liquid-biopsy guided Intensive Surveillance arm for whom a via imaging verified recurrence is documented during the 5-year interventional period of the study. If a patient has a via imaging verified recurrence but no documented molecular relapse, the Lead Time for this patient is set to '0'. This secondary endpoint will be assessed for all markers in combination and, where applicable, for each marker separately.
Quality of life (QoL) with questionnaires: EORTC QLQ-C30 | 10 years
  QoL will be monitored in both groups using a questionnaire which is to be completed every 6 months (EORTC QLQ-C30) in the interventional phase (first five years) and once a year during the five years of follow-up. QoL data will be collected on paper or via a digital health application.
Quality of life (QoL) with questionnaires: PA-F12 | 10 years
  QoL will be monitored in both groups using a questionnaire which is to be completed every 6 months (PA-F12) in the interventional phase (first five years) and once a year during the five years of follow-up. QoL data will be collected on paper or via a digital health application.
Liquid biopsy sensitivity (CA27.29, CEA, CA125, CTC and ctDNA) | 5 years
  Sensitivity is defined as the proportion of all patients in the liquid-biopsy guided Intensive Surveillance arm with a recurrence as verified by imaging during the 5-year interventional period of the study that had a positive biomarker result (i.e., molecular relapse) within 36 months before the recurrence as verified by imaging occurred (or within 60 months before the recurrence as verified by imaging occurred if in the first 36 months at least once a year a positive biomarker is measured).
Liquid biopsy specificity (CA27.29, CEA, CA125, CTC and ctDNA) | 5 years
  Specificity is defined as the proportion of all patients in the liquid-biopsy guided Intensive Surveillance arm with no recurrence as verified by imaging during the 5-year interventional period of the study that had only negative biomarker results (i.e., no indication of molecular relapse) within 36 months before the end of the 5-year interventional period of the study.
Liquid Biopsy False-Positive Rate (CA27.29, CEA, CA125, CTC and ctDNA) | 5 years
  False-positive rate is defined as the proportion of all patients in the liquid-biopsy guided Intensive Surveillance arm with a positive biomarker result (i.e., molecular relapse) during the 5-year interventional period of the study that had no recurrence as verified by imaging within 36 months after first molecular relapse.
Liquid Biopsy False-Negative Rate (CA27.29, CEA, CA125, CTC and ctDNA) | 5 years
  False-negative rate is defined as the proportion of all patients in the liquid-biopsy guided Intensive Surveillance arm with only negative biomarker results (i.e., no indication of molecular relapse) that had a recurrence as verified by imaging during the 5-year interventional period of the study.
Rate of liquid biopsy positivity (CA27.29, CEA, CA125, CTC and ctDNA) | 5 years
  The overall rate of liquid biopsy positivity is defined as the proportion of all patients in the liquid-biopsy guided Intensive Surveillance arm that had at least one positive biomarker result (i.e., molecular relapse) during the 5-year interventional period of the study.

OTHER OUTCOMES:
Establishment of a Biobank for Translational Research Endpoint | 5 years
  A biobank will allow the storage of unused biomaterials from both, the Intensive Surveillance arm as well as the Standard Surveillance arm. These materials will be used for future retrospective studies.

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Huesmann, Dr., Principal Investigator — Universitätsklinikum Ulm
Locations (1):
- University Hospital Ulm Gynecology/Obstetrics, Ulm, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://www.survive-studie.de

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-02): https://cdn.clinicaltrials.gov/large-docs/72/NCT05658172/Prot_SAP_000.pdf